CLINICAL TRIAL: NCT02326077
Title: Intrapartum Ultrasonography - Sonopartogram. Longitudinal Evaluation of the Mechanism of Active Labor Using Ultrasound Parameters
Brief Title: Sonopartogram. The Next Step in the Delivery Room
Acronym: SONOLABOR
Status: Suspended | Type: Observational
Why Stopped: Equipment and personnel discontinuity
Sponsor: University of Medicine and Pharmacy Craiova (Other)
Collaborators: University of Athens (Other)
Responsible Party: Sponsor
Other Study IDs: SONOPARTOGRAM
Record Dates: First submitted 2014-12-20; First posted 2014-12-25 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Normal Labor; Obstetric Labor Complications
Keywords: sonopartogram; transperineal ultrasound; intrapartum ultrasound; labor; delivery; partogram; ultrasound
MeSH Terms: conditions — Obstetric Labor Complications | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intervention group: Clinical evaluation in active labor: Leopold manoeuvres, vaginal digital examination.
  Transabdominal and transperineal ultrasound evaluations of the mechanism of labor: fetal head position, progression and rotation.
  Investigation by questionnaire regarding the psychological impact of labor monitoring assisted by sonoraphy.
  Interventions: Other: Ultrasound; Other: Acceptability of ultrasound monitoring of labor; Other: Patients' experience regarding intrapartum ultrasound

INTERVENTIONS:
Other: Ultrasound — Monitoring of the mechanism of labor
Other: Acceptability of ultrasound monitoring of labor — Evaluation of the acceptability of intrapartum ultrasound monitoring - the rate of uptake ultrasound protocol during labor
Other: Patients' experience regarding intrapartum ultrasound — The day after birth, consenting women are invited to take part in a questionnaire survey. Questionnaires contained no identifying information other than a code number and contains features regarding the patient's impression about the ultrasound monitoring scans during labor. The final questions concerned the willingness of having again another such protocol for labor monitoring in the future.

SUMMARY:
Objectives:

* Evaluation of the correlation between the sonographic parameter and clinical findings (e.g. digital examination) in any cephalic (not only occipital anterior) position
* Examination of the relationship between various sonographic parameters
* Determination of intraobserver and interobserver variation in obtaining the sonographic measurements
* Analysis of the temporal variation of the different sonographic measurements in normal spontaneous vaginal delivery versus obstructed labor in fetuses with occiput anterior versus those with persistent occiput posterior
* Establishment of a sonopartogram that should replace in an objective way Friedmann
* Establishment of cut-off values that may help clinicians to choose between vaginal operative delivery or caesarean section
* Another interesting aspect of intrapartum transperineal ultrasound imaging is whether there is a psychological benefit to the patient in being able to follow on the ultrasound screen how fetal head descent and position are being assessed objectively.

DETAILED DESCRIPTION:
Objectives:

* Evaluation of the correlation between the sonographic parameter and clinical findings (e.g. digital examination) in any cephalic (not only occipital anterior)
* Examination of the relationship between various sonographic parameters
* Determination of intraobserver and interobserver variation in obtaining the sonographic measurements
* Analysis of the temporal variation of the different sonographic measurements in normal spontaneous vaginal delivery versus obstructed labor in fetuses with occiput anterior versus those with persistent occiput posterior
* Establishment of a sonopartogram that should replace in an objective way Friedmann
* Determination of cut-off values that may help clinicians to choose between vaginal operative delivery or caesarean section
* Investigation whether there is a psychological benefit to the patient in being able to follow on the ultrasound screen how fetal head descent and position are being assessed objectively.

Methods:

Unselected population Personal characteristics: GA, BMI, age, gesta, para Gestational age of more than 37 completed weeks dated by first- and/or mid-trimester scan.

Each patient provide informed consent before the ultrasound measurements. Transperineal ultrasound imaging and digital examinations in laboring patients with a singleton fetus in cephalic/pelvic presentation. Patients examined in their labor rooms.

Admission time:

* active labor demonstrated by regular uterine contractions and changes in cervical dilatation of more than 2 cm,
* subgroup: prolonged second stage of labor (full cervical dilatation for >3 h if regional anesthesia was administered or 2 h in the absence of regional anesthesia in nulliparous women, or for >2 h with regional anesthesia or 1 h without anesthesia in parous women).

Empty bladder. Ultrasound machine with a 3.5-5MHz transducer used for the TA and TPU measurements. The probe enclosed in a latex glove covered with ultrasound gel and was then placed between the labia below the pubic symphysis/perineal.

Measured parameters:

Clinical examination (digital vaginal + Leopold) followed immediately after by the acquisition of the sonographic planes necessary to evaluate:occiput position, the long axis of the pubic symphysis, the infrapubic line, the progression angle, the distance of progession, the direction of progression, the midline angle, the head to perineum distance.

Identification and measurement of caput succedaneum (vertical+orizontal) and molding (vertical) when present.

All parameters recorded electronically for later analysis + volumes, when possible.

TPU scans performed at different times during labor,

* Hourly until complete dilation (1st phase)
* At 10 minutes after complete dilation (2nd phase) (at least one contraction between the examinations).

Notation of time delivery later used to calculate the interval from scanning to delivery.

In all cases measurements are performed in concert with digital examinations (immediately after).

Intraobserver and interobserver analysis 100 women assessed by TPU examination in the study, have at least one set of two replicated scans obtained at approximately the same time. These women provide sets of scans at various times throughout labor, used to assess intraobserver variability.

In order to assess interobserver variability, a second/independent and well trained observer, blinded to the other's results,

* obtain duplicate sets of scans at distinct times of labor among randomly selected women (one woman repeated at three time points). The consecutive scans performed with no more than 3 min between the assessments of the two observers
* or measuring the parameters stored on 3D volumes by the first observer The goal is to generate paired sets of replicated images under nearly identical conditions.

The measurements from the ultrasound scanning are obtained offline, after the acquisition of the described planes, on the images stored on the US machine hard disk.

Thus, the managing obstetrician is blinded to the transperineal ultrasound findings. Head position obtained by ultrasound imaging is communicated in case of clinical misdiagnose because of ethical reasons.

The decision whether expectant management, vaginal extraction or Cesarean section is appropriate is made exclusively on the basis of clinical examination.

Demographic data are collected including length of the second stage of labor, mode of delivery, maternal and neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* active labor
* singleton pregnancy
* eutrophic fetus
* cephalic presentation

Exclusion Criteria:

* indication for elective caesarean section
* non-cephalic presentation
* prior caesarean delivery
* fetal hypotrophy or macrosomy
* multiple pregnancies

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The pregnant women admitted in active labor at term were considered eligible for the study.
  They are included in the study consecutively, depending on the availability of the US operators involved.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Sonopartogram. Longitudinal assessment of the mechanism of labor using ultrasound parameters. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicolae Cernea, Professor, Study Chair — University of Medicine and Pharmacy Craiova; Dominic G Iliescu, Lecturer, Study Director — University of Medicine and Pharmacy Craiova; Stefania Tudorache, Lecturer, Principal Investigator — University of Medicine and Pharmacy Craiova
Locations (2):
- Alexandra University Hospital, Athens, Greece
- University Emergency County Hospital, Craiova, Dolj, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang J, Troendle JF, Yancey MK. Reassessing the labor curve in nulliparous women. Am J Obstet Gynecol. 2002 Oct;187(4):824-8. doi: 10.1067/mob.2002.127142. PMID 12388957
- [Background] Rayburn WF, Siemers KH, Legino LJ, Nabity MR, Anderson JC, Patil KD. Dystocia in late labor: determining fetal position by clinical and ultrasonic techniques. Am J Perinatol. 1989 Jul;6(3):316-9. doi: 10.1055/s-2007-999602. PMID 2659012
- [Background] Kreiser D, Schiff E, Lipitz S, Kayam Z, Avraham A, Achiron R. Determination of fetal occiput position by ultrasound during the second stage of labor. J Matern Fetal Med. 2001 Aug;10(4):283-6. doi: 10.1080/714904341. PMID 11531156
- [Background] Sherer DM, Miodovnik M, Bradley KS, Langer O. Intrapartum fetal head position I: comparison between transvaginal digital examination and transabdominal ultrasound assessment during the active stage of labor. Ultrasound Obstet Gynecol. 2002 Mar;19(3):258-63. doi: 10.1046/j.1469-0705.2002.00641.x. PMID 11896947
- [Background] Sherer DM, Miodovnik M, Bradley KS, Langer O. Intrapartum fetal head position II: comparison between transvaginal digital examination and transabdominal ultrasound assessment during the second stage of labor. Ultrasound Obstet Gynecol. 2002 Mar;19(3):264-8. doi: 10.1046/j.1469-0705.2002.00656.x. PMID 11896948
- [Background] Akmal S, Tsoi E, Kametas N, Howard R, Nicolaides KH. Intrapartum sonography to determine fetal head position. J Matern Fetal Neonatal Med. 2002 Sep;12(3):172-7. doi: 10.1080/jmf.12.3.172.177. PMID 12530614
- [Background] Souka AP, Haritos T, Basayiannis K, Noikokyri N, Antsaklis A. Intrapartum ultrasound for the examination of the fetal head position in normal and obstructed labor. J Matern Fetal Neonatal Med. 2003 Jan;13(1):59-63. doi: 10.1080/jmf.13.1.59.63. PMID 12710859
- [Background] Iliescu DG, Adam G, Tudorache S, Antsaklis P, Cernea N. Quantification of fetal head direction using transperineal ultrasound: an easier approach. Ultrasound Obstet Gynecol. 2012 Nov;40(5):607-8. doi: 10.1002/uog.11117. Epub 2012 Sep 24. No abstract available. PMID 22302748
- [Background] Hassan WA, Eggebo T, Ferguson M, Gillett A, Studd J, Pasupathy D, Lees CC. The sonopartogram: a novel method for recording progress of labor by ultrasound. Ultrasound Obstet Gynecol. 2014 Feb;43(2):189-94. doi: 10.1002/uog.13212. PMID 24105734
- [Background] Eggebo TM. Ultrasound is the future diagnostic tool in active labor. Ultrasound Obstet Gynecol. 2013 Apr;41(4):361-3. doi: 10.1002/uog.12417. No abstract available. PMID 23641509
- [Background] FRIEDMAN EA. Primigravid labor; a graphicostatistical analysis. Obstet Gynecol. 1955 Dec;6(6):567-89. doi: 10.1097/00006250-195512000-00001. No abstract available. PMID 13272981
- [Background] Tutschek B, Braun T, Chantraine F, Henrich W. A study of progress of labour using intrapartum translabial ultrasound, assessing head station, direction, and angle of descent. BJOG. 2011 Jan;118(1):62-9. doi: 10.1111/j.1471-0528.2010.02775.x. Epub 2010 Nov 18. PMID 21083864
- [Derived] Dira LM, Tudorache S, Antsaklis P, Daskalakis G, Themistoklis D, Belciug S, Stoean R, Novac M, Cara ML, Dragusin R, Florea M, Patru C, Zorila L, Nagy R, Ruican D, Iliescu DG. Sonographic Evaluation of the Mechanism of Active Labor (SonoLabor Study): observational study protocol regarding the implementation of the sonopartogram. BMJ Open. 2021 Sep 7;11(9):e047188. doi: 10.1136/bmjopen-2020-047188. PMID 34493509